CLINICAL TRIAL: NCT02064179
Title: Assessment of Efficacy of the First Aspirin Dose in Children Undergoing Surgery for Congenital Heart Disease (CHD) Who Require Post-operative Antiplatelet Therapy; Evaluated by Thromboelastograph (TEG) Analysis and TEG-platelet Mapping
Brief Title: Assessment of the Efficacy of the First Aspirin Dose in Children Undergoing Surgery for Congenital Heart Disease (CHD) Who Require Post-operative Antiplatelet Therapy
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-3167; UL1TR001082 (NIH)
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Antiplatelet therapy; Aspirin
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples for immediate processing via thromboelastograph (TEG) and TEG-platelet mapping (TEG-PM)
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of heparin and aspirin for their respective anticoagulation and antiplatelet effects is routine in intensive care units around the country and world in children who have undergone surgery for congenital heart disease (CHD) who are at risk for thrombosis after repair. Most common protocols recommend heparin infusions after surgery with transition to oral aspirin when oral intake begins. Patients at risk for thrombosis after congenital heart surgery requiring long-term antiplatelet therapy include those undergoing shunt placement for single-ventricle palliation or establishment of pulmonary blood flow, valve replacements, or coronary artery manipulation. Post-operative thrombosis after congenital heart surgery is rare, but thrombosis can result in death. The routine use of aspirin in these patients is intended to prevent the potentially catastrophic consequences of thrombosis. However, there is no routine clinical assessment of the platelet inhibitory effect of aspirin; nor have there been any prospective studies to assess the effectiveness of aspirin's antiplatelet effect in children after congenital heart surgery. No data exists to suggest that the first dose of aspirin transition from heparin infusion is either sufficient or insufficient in its antiplatelet effect.

In this study, the investigators will evaluate the effectiveness of the first aspirin dose in its antiplatelet effects after surgery for congenital heart disease. Degree of antiplatelet effect will be evaluated with thromboelastograph (TEG) and TEG-platelet mapping study analysis. Thromboelastography is a clinical laboratory method of assessing whole blood hemostasis and allows for assessment of clot formation, strength, and stability. TEG is most commonly used in patients at risk for bleeding or thrombosis and also to monitor antiplatelet therapies (such as aspirin).

The investigators hypothesize: the first dose of aspirin transitioned from heparin infusion after congenital heart surgery is sufficient in its antiplatelet effect as tested by TEG and TEG-platelet mapping studies. Confirmation of the antiplatelet effect of aspirin will help support the current practice of empiric aspirin therapy to prevent post-operative thrombosis in children after congenital heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18
* Undergoing surgery for congenital heart disease requiring oral antiplatelet therapy

Exclusion Criteria:

* Strict: personal or family history of bleeding/clotting disorder, patients requiring anticoagulation rather than antiplatelet therapy after surgery.
* Relative: patients with significant post-operative bleeding precluding the use of anticoagulation and/or antiplatelet therapy within the first 48-72 hours (eg. clinical instability preventing the initiation of oral aspirin therapy), patients requiring additional fresh platelet transfusion after the initiation of post-operative heparin infusion.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes children aged 0-18 with congenital heart disease (CHD) in the immediate post- operative period who receive heparin infusion prior to initiation of long-term antiplatelet therapy. The current study population includes patients who have undergone one of these surgeries requiring aspirin therapy. The following are the surgical procedures included in this study:
  1. Arterio-venous shunts: classic and modified Blalock-Taussig (BT) shunts, and central shunts.
  2. Veno-venous shunts: partial cavo-pulmonary connections (Glenn anastomosis), total cavo-pulmonary shunts (Fontan), and right ventricle to pulmonary artery conduits.
  3. Patients requiring coronary artery re-implantation: arterial switch operation for transposition of the great arteries and repair of anomalous left coronary artery arising from the pulmonary artery.
  4. Pulmonary valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Full platelet inhibition with aspirin 4-hours after surgery compared to prior to surgery | 4-hours after first aspirin dose
  We will obtain thromboelastograph and thromboelastograph-platelet mapping studies at 4 time points: (1) prior to surgery and cardiopulmonary bypass, (2) 24-hours prior to the first aspirin dose, (3) 4-hours after the first aspirin dose, (4) 24-hours after the first aspirin dose (prior to the second).
  Primary Outcome measure will compare the first-postoperative TEG/TEG-platelet mapping results (4-hours after surgery) to the pre-operative TEG/TEG-platelet mapping results (prior to surgery)

SECONDARY OUTCOMES:
Full platelet inhibition at 24-hours if not achieved by 4-hours after aspirin administration | 24-hours after first aspirin dose (prior to second)
  We will obtain thromboelastograph and thromboelastograph-platelet mapping studies at 4 time points: (1) prior to surgery and cardiopulmonary bypass, (2) 24-hours prior to the first aspirin dose, (3) 4-hours after the first aspirin dose, (4) 24-hours after the first aspirin dose (prior to the second).
  Secondary outcome will compare 24-hour TEG/TEG-platelet mapping to 4-hour TEG/TEG-platelet mapping after surgery